CLINICAL TRIAL: NCT06677983
Title: Clinical Performance and Acceptance of Bioflx Crowns: a Randomized Controlled Clinical Trial
Brief Title: Clinical Performance and Acceptance of Bioflx Crowns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02202409293266
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioflex (Experimental)
  Interventions: Other: Bioflex Crowns
- SSC (Active Comparator)
  Interventions: Other: Stainless steel crown

INTERVENTIONS:
Other: Bioflex Crowns — A preformed crown of similar size will be selected. Tooth preparation will be done using a tapered diamond bur to reduce the occlusal surface, including the central groove, by 1-1.5 mm. The proximal surfaces will be prepared by approximately 0.5 mm to clear the contact area.
  Arms: Bioflex
Other: Stainless steel crown — An appropriately sized preformed stainless-steel crown will be selected. Tooth preparation will involve using a tapered bur ) to reduce the occlusal surface by 1 to 1.5 mm, with interproximal reduction made on the mesial and distal sides. The selected crown size will be checked, and a trial fit will be conducted prior to cementation. Crimping pliers will be used, and the crown will be cemented with Type 1 glass ionomer cement. Any excess cement will be removed, and proper occlusion will be verified.
  Arms: SSC

SUMMARY:
Treating pediatric patients with early childhood caries can be challenging. For clinicians, managing a young child while ensuring high-quality treatment is difficult. It is essential to have the best equipment and materials available. Today, aesthetics are crucial in managing decayed teeth, with zirconia crowns often preferred for their visual appeal, although they require substantial preparation. The newly developed Bioflx crown, combining stainless steel and zirconia properties, offers an alternative solution.

ELIGIBILITY:
Inclusion Criteria:

* A child with primary molars is indicated for full coverage.

Exclusion Criteria:

* Children with any systemic disease
* Clinical or radiographic signs/symptoms of irreversible pulpitis as abscess, fistula, spontaneous pain, mobility, furcation involvement, internal or external root resorption
* Children cooperation (1,2) according to Frankl scale
* Parents are unwilling to enroll their children in study

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in clinical success | baseline, 6 months, and 12 months
  The crowns were evaluated clinically according to the following criteria: 1. Length: the margin is at the gingival crest or is extended to the cemento-enamel junction. 2. Position: crown is not rotated. 3. Polish: no scratches or roughness. 4. Cement: no excess cement remains in the sulcus. If all criteria fulfilled the crown is considered acceptable clinically, if not it is considered unacceptable.
parental satisfaction | through study completion, an average of 6 months
  The questionnaire for assessing parental satisfaction includes four main categories for rating the aesthetic characteristics: size, shape, color, and stain.
  Responses will be recorded on a five-point Likert scale, ranging from 1 (not at all satisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Pediatric dentistry, Faculty of dentistry, pharos University, Egypt, Alexandria, Egypt